CLINICAL TRIAL: NCT06321146
Title: Evaluation of EEG Power Spectrum in Patients With Traumatic Coma
Acronym: EPIC
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Xiangya Hospital of Central South University (Other); The General Hospital of Eastern Theater Command (Other); Anhui No.2 Provincial People's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: LY2024-029-B
Record Dates: First submitted 2024-03-10; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Coma; Brain Injuries, Traumatic
Keywords: Coma; Traumatic brain injury; EEG power spectrum
MeSH Terms: conditions — Coma; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- V-P shunt group: Comatose TBI patients who underwent V-P shunt surgery
- Cranioplasty group: Comatose TBI patients who underwent cranioplasty surgery
- SCS group: Comatose TBI patients who underwent spinal cord stimulation
- RMNS group: Comatose TBI patients who underwent right median nerve stimulation
- DAI group: Comatose TBI patients with diffuse axonal injury

SUMMARY:
Development of objective, reliable, and convenient assessment methods of disorders of consciousness is crucial. We aim to conduct multicenter prospective observational study and non-invasively collect EEG from patients with traumatic coma to analyze the sequential characteristics of EEG power spectrum, and explore their prognostic value for consciousness recovery.

DETAILED DESCRIPTION:
Trauma brain injury is a leading cause of chronic disorders of consciousness (DoC), posing significant socioeconomic burdens due to the extensive resources required for long-term medical care. DoC patients are clinically categorized into coma, Unresponsive Wakefulness Syndrome (UWS) and Minimally Conscious State (MCS), with the latter further subdivided into MCS- and MCS+. The Coma Recovery Scale-Revised (CRS-R) remains a cornerstone for diagnosis and assessment of DoC, despite its susceptibility to fluctuations caused by various factors such as comorbidities and medication. Given these challenges, the development of objective, reliable, and convenient assessment methods of DoC is crucial. Electroencephalography (EEG) stands out for its accessibility and is recommended by guidelines. The mesocircuit model underscores the role of central thalamic neurons and their frontostriatal connections in maintaining consciousness. Based on this mechanism, EEG power spectra were categorized into 4 patterns, i.e. the ABCD model, which can be used to understand the varying levels of structural or functional deafferentation that occur in patients with DoC. Preliminary studies have shown the potential of corticothalamic EEG classification in correlating with CRS-R scores and neurological outcomes, suggesting its value in monitoring treatment effects and predicting prognosis. This multicenter prospective observational study aims to enroll patients with traumatic coma, analyze the sequential characteristics of corticothalamic EEG power spectrum, and explore their prognostic value for consciousness recovery.

ELIGIBILITY:
Inclusion Criteria:

* Coma over 28 days due to closed traumatic brain injury
* Age above 18 years old
* Consented by legal representative

Exclusion Criteria:

* Unstable vital signs
* History of mental disorder or neurodegenerative diseases
* Uncontrolled epilepsy
* Unable to record scalp EEG
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with traumatic coma above 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
EEG power spectrum | within 6 months after discharge
  Sequential characteristics of spectral features for EEG in terms of frequency content (the 'ABCD' spectral categories)

SECONDARY OUTCOMES:
Coma Recovery Scale-Revised (CRS-R) | within 6 months after discharge
  Coma Recovery Scale-Revised in patients with traumatic coma

CONTACTS AND LOCATIONS:
Overall Officials: Junfeng Feng, Dr., Study Director — Renji Hospital, School of Medicine, Shanghai Jiaotong University; Guoyi Gao, Dr., Study Director — Beijing Tiantan Hospital; Jinfang Liu, Dr., Study Director — Xiangya Hospital of Central South University; Chiyuan Ma, Dr., Study Director — The General Hospital of Eastern Theater Command; Yongming Zhang, Dr., Study Director — Anhui No.2 Provincial People's Hospital
Locations (5):
- China (5):
  - Anhui No.2 Provincial People's Hospital, Hefei, Anhui
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - The General Hospital of Eastern Theater Command, Nanjing, Jiangsu
  - Brain Injury Center, Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
Researchers who submit a methodologically sound study proposal that is approved by the management committee can have access to the study protocol, individual participant data and data dictionary. A Data Access Agreement is required, and all access must comply with regulatory restrictions imposed on the original study.
Supporting Information: Study Protocol
Time Frame: After Publication
Access Criteria: Researchers who submit a methodologically sound study proposal that is approved by the management committee can have access to the study protocol, individual participant data and data dictionary.

REFERENCES:
- [Background] Edlow BL, Claassen J, Schiff ND, Greer DM. Recovery from disorders of consciousness: mechanisms, prognosis and emerging therapies. Nat Rev Neurol. 2021 Mar;17(3):135-156. doi: 10.1038/s41582-020-00428-x. Epub 2020 Dec 14. PMID 33318675
- [Background] Schiff ND. Mesocircuit mechanisms in the diagnosis and treatment of disorders of consciousness. Presse Med. 2023 Jun;52(2):104161. doi: 10.1016/j.lpm.2022.104161. Epub 2022 Dec 20. PMID 36563999
- [Background] Forgacs PB, Frey HP, Velazquez A, Thompson S, Brodie D, Moitra V, Rabani L, Park S, Agarwal S, Falo MC, Schiff ND, Claassen J. Dynamic regimes of neocortical activity linked to corticothalamic integrity correlate with outcomes in acute anoxic brain injury after cardiac arrest. Ann Clin Transl Neurol. 2017 Jan 6;4(2):119-129. doi: 10.1002/acn3.385. eCollection 2017 Feb. PMID 28168211
- [Background] Comanducci A, Boly M, Claassen J, De Lucia M, Gibson RM, Juan E, Laureys S, Naccache L, Owen AM, Rosanova M, Rossetti AO, Schnakers C, Sitt JD, Schiff ND, Massimini M. Clinical and advanced neurophysiology in the prognostic and diagnostic evaluation of disorders of consciousness: review of an IFCN-endorsed expert group. Clin Neurophysiol. 2020 Nov;131(11):2736-2765. doi: 10.1016/j.clinph.2020.07.015. Epub 2020 Aug 14. PMID 32917521
- [Background] Thibaut A, Schiff N, Giacino J, Laureys S, Gosseries O. Therapeutic interventions in patients with prolonged disorders of consciousness. Lancet Neurol. 2019 Jun;18(6):600-614. doi: 10.1016/S1474-4422(19)30031-6. Epub 2019 Apr 16. PMID 31003899
- [Background] Alkhachroum A, Eliseyev A, Der-Nigoghossian CA, Rubinos C, Kromm JA, Mathews E, Bauerschmidt A, Doyle K, Velasquez A, Egbebike JA, Calderon AR, Roh DJ, Park S, Agarwal S, Connolly ES, Claassen J. EEG to detect early recovery of consciousness in amantadine-treated acute brain injury patients. J Neurol Neurosurg Psychiatry. 2020 Jun;91(6):675-676. doi: 10.1136/jnnp-2019-322645. Epub 2020 Apr 2. No abstract available. PMID 32241920
- [Background] Curley WH, Bodien YG, Zhou DW, Conte MM, Foulkes AS, Giacino JT, Victor JD, Schiff ND, Edlow BL. Electrophysiological correlates of thalamocortical function in acute severe traumatic brain injury. Cortex. 2022 Jul;152:136-152. doi: 10.1016/j.cortex.2022.04.007. Epub 2022 Apr 15. PMID 35569326
- [Background] Frohlich J, Crone JS, Johnson MA, Lutkenhoff ES, Spivak NM, Dell'Italia J, Hipp JF, Shrestha V, Ruiz Tejeda JE, Real C, Vespa PM, Monti MM. Neural oscillations track recovery of consciousness in acute traumatic brain injury patients. Hum Brain Mapp. 2022 Apr 15;43(6):1804-1820. doi: 10.1002/hbm.25725. Epub 2022 Jan 25. PMID 35076993